CLINICAL TRIAL: NCT05604014
Title: Feasibility Study of the My Health Coach App for Adults With Fetal Alcohol Spectrum Disorders (FASD)
Brief Title: Feasibility Study of the My Health Coach App for Adults With FASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christie Petrenko, Research Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00007749; UH2AA029050 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Health Coach (Experimental): Participants receive the My Health Coach app and try it on their personal smartphones for 6 weeks.
  Interventions: Behavioral: My Health Coach

INTERVENTIONS:
Behavioral: My Health Coach — My Health Coach is a self-directed mobile health intervention for adults with FASD. It is grounded in self-determination theory and integrates well-established behavior change strategies. It has a cloud-based infrastructure and uses a just-in-time adaptive intervention design and a simple and engaging chatbot interface. It provides adults just the right type and amount of support, when they are most receptive.

SUMMARY:
The purpose of this study is to test a new smartphone "app" for adults with fetal alcohol spectrum disorder (FASD). The app is called My Health Coach. The goal of the app is to provide adults with useful information and tools to help manage their health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older
* Have a fetal alcohol spectrum disorder (FASD) or history of prenatal alcohol exposure
* Have conversational fluency in English
* Own an smartphone

Exclusion Criteria:

* Unable to complete measures or interviews in English
* Do not have a smartphone
* Under 18
* Do not have an FASD or history or prenatal alcohol exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mt. Hope Family Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be deposited within the Collaborative Initiative on FASD (CIFASD) Central Repository and the National Institute on Alcohol Abuse and Alcoholism Data Archive as required by grant regulations. CIFASD Data Sharing policies and data access request information can be found at: https://cifasd.org/data-sharing/. NIAAA-DA access can be found at: https://nda.nih.gov/niaaa/
Supporting Information: Study Protocol, ICF
Time Frame: All collection data are shared automatically two years after the grant end date.
Access Criteria: See https://nda.nih.gov/niaaa/ for details.
URL: https://nda.nih.gov/niaaa/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 95 enrolled in the study, 52 were excluded for the following reasons: 2 did not meet eligibility criteria, 1 declined to participate, 5 had incomplete screening data, 7 were duplicates, and 37 were suspected fraudulent participants.
Period: Overall Study
Arm/Group | My Health Coach
Started | 43
Baseline Surveys | 39
Installed App | 33
6-Week Follow-up Surveys | 30
Completed | 30
Not Completed | 13
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | My Health Coach
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 29
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
  Canada | 7
  Netherlands | 4
  United Kingdom | 4
  Ireland | 1
  Italy | 1
  New Zealand | 1
  South Africa | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Subjective Well-being From Baseline to 6-week Follow-up on the Personal Well-Being Index - Intellectual Disability Version
Description: The Personal Well-Being Index (PWI) is an 7-item measure of subjective well-being. The Intellectual Disability Version uses more concrete item wording and a 5-point visual scale. Ratings are averaged and the mean total is reported ranging from 1 to 5. Higher scores reflect better perceived well-being.
Time Frame: Baseline to 6 Weeks
Population: Participants with complete data at baseline and 6-week follow-up surveys are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | My Health Coach
Number analyzed (Participants) | 30
units on a scale
  Baseline | 3.51 (0.68)
  6-Week Follow-up | 3.59 (0.69)
Statistical Analysis 1: Comparison: My Health Coach; Test type: Superiority; p = 0.49, t-test, 2 sided; Mean Difference (Final Values) = -0.7

2. Primary Outcome: Mean Change in Autonomy Ratings From Baseline to 6-week Follow-up on the Basic Psychological Need Satisfaction and Frustration Scale - Autonomy Sub-scale
Description: The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSF) is a 24-item scale assessing both satisfaction and frustration relating to the three basic psychological needs identified in self-determination theory: autonomy, competence, and relatedness. Items are rated on a 5-point scale from 1 "not at all true" to 5 "completely true." Each sub-scale has 8 items. Scores were averaged across items with reported mean ranging from 1 to 5. Higher scores reflect higher satisfaction or need being met to a higher degree. The Autonomy sub-scale measures how much a person feels they have choice in what they do in their everyday life.
Time Frame: Baseline to 6 Weeks
Population: Participants with completed data at both baseline and 6-week follow-up timepoints were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | My Health Coach
Number analyzed (Participants) | 28
units on a scale
  Baseline | 3.38 (0.59)
  6-Week follow-up | 3.46 (0.49)
Statistical Analysis 1: Comparison: My Health Coach; Test type: Superiority; p = 0.5, t-test, 2 sided; Mean Difference (Final Values) = -0.69

3. Primary Outcome: Mean Change in Competence Ratings From Baseline to 6-week Follow-up on the Basic Psychological Need Satisfaction and Frustration Scale - Competence Sub-scale
Description: The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSF) is a 24-item scale assessing both satisfaction and frustration relating to the three basic psychological needs identified in self-determination theory: autonomy, competence, and relatedness. Items are rated on a 5-point scale from 1 "not at all true" to 5 "completely true." Each sub-scale has 8 items. Scores were averaged across items with reported mean ranging from 1 to 5. Higher scores reflect higher satisfaction or need being met to a higher degree. The Competence sub-scale measures how much a person feels they are successful or do a good job on things in their life.
Time Frame: Baseline to 6 Weeks
Population: Participants with complete data at both baseline and 6-week follow-up timepoints were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | My Health Coach
Number analyzed (Participants) | 28
units on a scale
  Baseline | 3.12 (0.67)
  6-week follow-up | 3.32 (0.5)
Statistical Analysis 1: Comparison: My Health Coach; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = -1.44

4. Primary Outcome: Mean Change in Relatedness Ratings From Baseline to 6-week Follow-up on the Basic Psychological Need Satisfaction and Frustration Scale - Relatedness Sub-scale
Description: The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSF) is a 24-item scale assessing both satisfaction and frustration relating to the three basic psychological needs identified in self-determination theory: autonomy, competence, and relatedness. Items are rated on a 5-point scale from 1 "not at all true" to 5 "completely true." Each sub-scale has 8 items. Scores were averaged across items with reported mean ranging from 1 to 5. Higher scores reflect higher satisfaction or need being met to a higher degree. The Relatedness sub-scale measures how much a person feels connected to other people in their life.
Time Frame: Baseline to 6 Weeks
Population: Participants with completed data at both baseline and 6-week follow-up timepoints were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | My Health Coach
Number analyzed (Participants) | 28
units on a scale
  Baseline | 3.48 (0.69)
  6-week Follow-up | 3.58 (0.58)
Statistical Analysis 1: Comparison: My Health Coach; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = -0.78

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events in adults with FASD could include aggression or violence towards others, self-harm or suicidality, or the need for inpatient hospitalization. However, these occurrences are unlikely to be a direct consequence of participation in the app intervention or study. These were not systematically assessed but procedures were in place to assess risk and respond appropriately if they arose.
Arm/Group | My Health Coach
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT05604014/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT05604014/ICF_001.pdf